CLINICAL TRIAL: NCT06297876
Title: COVIDVaxStories: A Pilot Double-blind Randomized, Parallel Design Trial of Storytelling to Reduce COVID-19 Vaccine Hesitation in Populations of Color Using a Respondent-driven Sampling Design
Brief Title: COVIDVaxStories: Randomized Trial to Reduce COVID-19 Vaccine Hesitancy in Populations of Color
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Jeroan Allison, Chair, Population and Quantitative Health Sciences, University of Massachusetts, Worcester
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: H00023815
Record Dates: First submitted 2023-05-01; First posted 2024-03-07 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Vaccine Hesitancy
MeSH Terms: conditions — Vaccination Hesitancy | interventions — Narrative Therapy

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will view either storytelling videos or learn more videos. They will not know which video they will get ahead of time nor will they know that they may get one or the other.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Storytelling (Experimental): Participants will view short video narratives of community members speaking about why they chose to get vaccinated against Coronavirus Disease of 2019 (COVID-19) and how they overcame hesitancy. Participants will also view the informational videos described below.
  Interventions: Behavioral: Storytelling
- Learn More (Other): Participants will view short informational videos that provide factual information on the COVID-19 vaccines.
  Interventions: Behavioral: Learn More (Active Comparator)

INTERVENTIONS:
Behavioral: Storytelling — Narrative stories will be videos that are 2-3 minutes long and will show community members speaking based on community identified themes.
  Other Names: Narrative
  Arms: Storytelling
Behavioral: Learn More (Active Comparator) — Informational videos that are of similar length and on the same topic as the storytelling videos.
  Arms: Learn More

SUMMARY:
Pilot randomized controlled trial testing the investigator's previously developed storytelling method to create an interactive, multi-media storytelling intervention to address community-identified reasons for vaccine hesitancy among Black and Hispanic individuals in Central Massachusetts

DETAILED DESCRIPTION:
Intervention Development The investigators will recruit 64-80 Black and Hispanic community members for storytelling development groups (described below) through our already established COVID community advisory board (C-CAB). The C-CAB represents ten community organizations throughout the Greater Worcester area including churches and community centers. Further information on procedures for intervention development can be found in the "study procedures" section.

Pilot Randomized Controlled Trial (RCT) The investigators will conduct a pilot feasibility randomized controlled trial. The investigators will enroll approximately 50 Black persons who identify as Black and/or Hispanic in Central Massachusetts. The investigators will use a Respondent-Driven Sampling (RDS) Design, a quantitative form of the "snowballing" approach that has been proven effective in under-represented groups19-22 to pilot our recruitment strategy. In RDS a preset number of "seeds" are selected with the assistance of community partners. The seeds are community members with large social networks. Each seed recruits a preset number of participants utilizing their social networks and this process continues in waves until the predetermined sample size is met. Each seed is linked to their recruits to enable social network analysis.

Study procedures from consent to intervention will be delivered through Qualtrics, an online service that allows researchers to design and deliver online research instruments with minimal time and effort, and without extensive programming experience (Qualtrics.com). A short screening survey, e-informed-consent form, surveys, and videos (both English and Spanish versions) will be uploaded into Qualtrics. Qualtrics is available on both mobile devices and desktops,14 through mobile app or internet. The University of Massachusetts Chan Medical School (UMMS) has a university license to use Qualtrics, which provide robust data safety and privacy and is approved by our Institutional Review Board (IRB). The investigators will utilize the Quantitative Methods Core (QMC), a service core that has been formed under the auspices of the Division of Biostatistics and Health Services Research within the Department of Population and Health Sciences as well as our current research coordinator who have partnered to create a Qualtrics interface that delivers pre-intervention surveys, randomization, intervention delivery, and post intervention surveys, for our completed Enhancing racial and ethnic diversity in COVID-19 research participation through storytelling (COVIDstory)study. Qualtrics has also previously been used for the aforementioned features for an intervention aimed at increasing uptake of the Human Papillomavirus (HPV) vaccine among young Asian women.14 The investigators will build on this infrastructure to tailor the randomization, surveys, and intervention delivery for this intervention in this population.

Participants will be randomly assigned to either the storytelling arm or the comparison arm through a randomization algorithm embedded within Qualtrics. A stratified approach will be used, with equal enrollment by racial/ethnic category: Black or Hispanic. Each person recruited will be directed to Qualtrics which will be set to proceed in a systematic and sequential manner until the full sample size of 25 participants in the intervention group and 25 participants in the comparison group, stratified by race/ethnicity, are attained. Study subjects and investigators will be blinded as to group assignment. As with our current NCI funded project, all participant-facing aspects of Qualtrics (screening, consent, randomization, surveys, intervention videos) will be available in both English and Spanish. .

ELIGIBILITY:
Inclusion Criteria:

* >= 18 years of age
* identifies as Black and/or Hispanic
* lives in Massachusetts
* vaccinated for COVID-19.

Exclusion Criteria:

* Unable to provide consent in English or Spanish
* Has not completed the primary series of COVID-19 vaccinations (2 shots for Moderna or Pfizer, one shot for Johnson & Johnson).

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-05-19 (Actual); Primary Completion 2024-08-09 (Actual); Study Completion 2024-08-09 (Actual)

PRIMARY OUTCOMES:
Change in Vaccine Hesitancy | From beginning of survey to end of survey typically, 30 minutes
  Validated vaccine hesitancy questionnaire

SECONDARY OUTCOMES:
Vaccine Uptake | 6 months after participation
  Percent in each study arm whose vaccination status changed post intervention by querying the participant. The investigators will also pilot test their willingness to provide the investigators with proof of vaccination (e.g., documentation from vaccinating entity or excerpt from electronic health record, if a change is reported

CONTACTS AND LOCATIONS:
Locations (1):
- University of Massachusetts Chan Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No